CLINICAL TRIAL: NCT05838404
Title: M-O-M-S on the Bayou: Implementation of an Intervention for Mental Health in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-1533
Record Dates: First submitted 2023-04-10; First posted 2023-05-01 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Depression
Keywords: Pregnancy; Pregnancy-related anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOMS on the Bayou Intervention Group (Experimental): Participants complete intervention protocol.
  Interventions: Behavioral: M-O-M-S on the Bayou

INTERVENTIONS:
Behavioral: M-O-M-S on the Bayou — Peer and mentor support and meetings across pregnancy

SUMMARY:
Disasters have negative effects in the short term (physical trauma, adverse environmental exposures, and unstable housing) and the long term (relocation, changes in family functioning, and negative economic effects), which interact with social determinants to worsen health among the most vulnerable women, infants, and communities. Trauma and severe stress are directly linked to pregnancy complications, and raise blood pressure during pregnancy, alter stress hormones, and increase vulnerability to infection, all of which predispose to reduced fetal growth and preterm birth. Disasters also worsen mental health, and depression during pregnancy and postpartum, for instance, is associated with worse physical health during pregnancy, maternal impairment, poorer quality parenting, negative child behavior, and poorer infant cognitive development.The goal of this intervention is to improve mental health in pregnant women living in a disaster-affected region.

The main questions this intervention aims to answer are:

* Assess the implementation outcomes (acceptability, adaptation, adoption, feasibility, fidelity, and sustainability) of a pilot intervention in a disaster recovery environment.
* Assess the effectiveness of the M-O-M-S pilot intervention in a disaster recovery environment.

The study will recruit pregnant women in areas that have experienced a natural disaster. Women will be recruited in early pregnancy and attend a series of classes on the cognitive and relationship changes of pregnancy and motherhood, and mental preparation for labor, led by a "mentor," a mother who has experienced pregnancy, labor, and motherhood.

DETAILED DESCRIPTION:
The M-O-M-S™ (Mentors Offering Maternal Support) intervention is based in a theoretical framework addressing the major transitions that occur with pregnancy and close relationship processes. Weis et al. found that community esteem-building support, focused in first and second trimester, decreased anxiety associated with pregnancy and maternal adaptation. The M-O-M-S™ intervention was specifically designed to address pregnancy-specific anxiety (inclusive of depressive symptoms), concerns related to family/partner relationships, and provide esteem-building peer support, with each session directly aligned to specific aspects of anxiety and depression pertinent to the point in pregnancy for the women. Women are recruited in early pregnancy and attend a series of classes on the cognitive and relationship changes of pregnancy and motherhood, and mental preparation for labor, led by a "mentor", a mother who has experienced pregnancy, labor, and motherhood.

Up to 400 subjects will be recruited, with a goal of 240 completing the study. Each group will consist of 15-20 recruits, assuming a degree of attrition that will lead to group sizes of 10-12. The outcome measures will be compared between the intervention and control data and linear regression (with adjustment for partial clustering) used to adjust for differences in participant characteristics. Given an estimated effect size and variance (both pre-post and intervention-control) from previous trials, 240 participants gives good power for reasonable effect sizes for both the pre-post analysis and intervention-control analyses incorporating a design (cluster) effect.

Recruitment will take place at ob/gyn practices, WIC clinics, health units, and at community sites. Clinicians will be informed of the intervention and asked to encourage their patients to participate. They will also refer potential participants and provide flyers to interested women. Study staff will also attend the clinics on days when a large number of prenatal visits are scheduled, and clinic staff will inform them who can be approached as a potential participant. Flyers and posters will also be provided to participating clinics, and participants can self-refer. Participants will be contacted via the method they indicate they prefer.

Participants will attend 6 group meetings lasting 1 hr. every other week. These sessions are aimed at decreasing pregnancy concerns and building coping skills through supportive relationships with experienced local mothers and the other participants in the group. The meetings are closed group sessions.

Participants also receive a "Birth of a Mother" manual designed to guide open discussion during the course of the sessions.

In addition, participants will complete questionnaires at baseline and at the end of the intervention about their mental health, experience of the intervention, and disaster experience.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Below 20 weeks' gestation
* Enrolled in prenatal care

Exclusion Criteria:

* Not pregnant
* Under age 18
* Does not speak English or Spanish
* Does not plan to carry to term
* Does not plan to remain in the study area through pregnancy
* Fetal defects likely to lead to death or extensive hospitalization postpartum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-specific anxiety | 12 weeks
  Score on the Lederman Prenatal Self-Evaluation Questionnaire (PSEQ), Scale of 1-4; 1 = worse outcome; 4 = better outcome.

SECONDARY OUTCOMES:
Depressive symptoms | 12 weeks
  Score on Edinburgh Postnatal Depression Scale (EPDS), Scale of 1-4; 1 = better outcome; 4 = worse outcome.

OTHER OUTCOMES:
Acceptability | 12 weeks
  Acceptability is assessed with the Acceptability of Intervention Measures (AIM) (Weiner BJ, Lewis CC, Stanick C, et. al.); Scale of 1-5; 1 = worse outcome; 5 = better outcome.
Fidelity | 12 weeks.
  Fidelity is measured as the number of sessions attended.

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from the intervention will be provided to the Gulf Research Program.
Time Frame: No later than two years after the end of the final participant follow-up or one year after the main paper of the project has been published, whichever comes first.
Access Criteria: Participant confidentiality is paramount and some topics (such as mental and reproductive health) are sensitive, so identifiers and any other data leading to possible deductive disclosure (such as small cell sizes) will be removed before provision to GRP.
URL: https://grp.griidc.org/